CLINICAL TRIAL: NCT00865774
Title: The Teachable Moment: Screening and Brief Intervention for Admitted Trauma Patients
Acronym: TM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00006734
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Alcoholism
Keywords: Trauma; Alcohol; Brief Intervention
MeSH Terms: conditions — Alcoholism; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Arm number 1 focuses on the traditional quantity frequency model.
  Interventions: Behavioral: Quantity Frequency Model
- 2 (Experimental): Arm number 2 targets subjective drunkenness.
  Interventions: Behavioral: Targets Subjective Drunkenness

INTERVENTIONS:
Behavioral: Quantity Frequency Model — The quantitative intervention involves emphasis on tracking and measuring the number of drinks on a weekly basis.
  Arms: 1
Behavioral: Targets Subjective Drunkenness — Explores factors leading to drunkenness and alternative coping strategies for healthier function.
  Arms: 2

SUMMARY:
The American College of Surgeons now requires screening for alcohol use in trauma centers. The purpose of this research study is to provide information about the best screening and treatment methods. The investigators hope the findings will provide information that will improve healthcare by reducing problems related to risky alcohol use. The trauma team is conducting a comparison of two different ways of talking about alcohol use. Participants will be randomized into one of the two study groups.

DETAILED DESCRIPTION:
The goal of this study is to guide further policy development regarding effective alcohol screening by: (a) comparing the effectiveness of two new, shorter screening tools for risky drinking patterns with the longer screening tool in current use; (b) assessing the outcomes of two different brief counseling interventions (BIs) with trauma patients screened to have risky drinking behaviors; and (c) examining the impact of the implementation of this new policy in a Level I Trauma Center.

The Specific Aims will be accomplished by:

1. Screening patients who are admitted to the Trauma Center, and conducting BIs for all who screen positive;
2. Collecting formative qualitative data regarding participants' perceptions of benefits of drunken states, their individual risks, and perceived healthier alternatives;
3. Collecting quantitative data (injury severity score and hospital length of stay) and correlating these data with patient demographics and responses on the different screening methods;
4. Collecting follow-up data by telephone on self-reported alcohol use and trauma recidivism, using an interviewer-administered assessment;
5. Collecting data on trauma recidivism from ED data, publicly available records, and patient self-report at 6-month telephone follow-up;
6. Surveying trauma staff and physicians at three intervals regarding the process of implementing the new ACS policy, any perceived difficulties, and the perceived impact

ELIGIBILITY:
Inclusion Criteria:

* Inpatient on trauma service
* 18 years or older
* Speaks either English or Spanish

One or more of the following:

* Patient answered yes to either admission screening question
* Patient has a positive BAL of less than or equal to 79 and also has a positive Audit score (men greater than or equal to 8; women greater than or equal to 4)
* Patient has a BAL of 80 or higher
* patient has no record of a BAL on file and they have a positive Audit score

Exclusion Criteria:

* Patient unable or unwilling to provide informed consent
* Patient refusal contact at six months
* Patient has a positive BAL of less than or equal to 79 and negative AUDIT score
* Patient deemed unable to complete a BI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Trauma recidivism after discharge as measured by a review of computerized ED records,NC Trauma database,the Forsyth County EMS registry,NC EMS registry and self-reports at a 6-month telephone follow-up of alcohol-related injuries and changes in alcohol | 6 months

SECONDARY OUTCOMES:
Patient satisfaction ratings of the BI,the response to the BI as rated by the interviewer,reported citations for driving under the influence(to be obtained from the NC State Department of Motor Vehicles) and 3 surveys of trauma service staff | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Claire O'Brien, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Fitzgerald DJ, Radek KA, Chaar M, Faunce DE, DiPietro LA, Kovacs EJ. Effects of acute ethanol exposure on the early inflammatory response after excisional injury. Alcohol Clin Exp Res. 2007 Feb;31(2):317-23. doi: 10.1111/j.1530-0277.2006.00307.x. PMID 17250625
- [Background] Zambell KL, Phelan H, Vande Stouwe C, Zhang P, Shellito JE, Molina PE. Acute alcohol intoxication during hemorrhagic shock: impact on host defense from infection. Alcohol Clin Exp Res. 2004 Apr;28(4):635-42. doi: 10.1097/01.alc.0000122104.85971.55. PMID 15100616
- [Background] Cunningham RM, Maio RF, Hill EM, Zink BJ. The effects of alcohol on head injury in the motor vehicle crash victim. Alcohol Alcohol. 2002 May-Jun;37(3):236-40. doi: 10.1093/alcalc/37.3.236. PMID 12003910
- [Background] Saitz R. Clinical practice. Unhealthy alcohol use. N Engl J Med. 2005 Feb 10;352(6):596-607. doi: 10.1056/NEJMcp042262. No abstract available. PMID 15703424
- [Background] National Highway Safety Traffic Administration. National Communications Plan 2006. http://www.nhtsa.dot.gov/people/injury/NewmediaForum Web/images/NHTS-1689%20Comm%20Plan.pdf Accessed March 18, 2008.
- [Background] Schermer CR, Moyers TB, Miller WR, Bloomfield LA. Trauma center brief interventions for alcohol disorders decrease subsequent driving under the influence arrests. J Trauma. 2006 Jan;60(1):29-34. doi: 10.1097/01.ta.0000199420.12322.5d. PMID 16456433
- [Background] Crawford MJ, Patton R, Touquet R, Drummond C, Byford S, Barrett B, Reece B, Brown A, Henry JA. Screening and referral for brief intervention of alcohol-misusing patients in an emergency department: a pragmatic randomised controlled trial. Lancet. 2004 Oct 9-15;364(9442):1334-9. doi: 10.1016/S0140-6736(04)17190-0. PMID 15474136
- [Background] Gentilello LM, Rivara FP, Donovan DM, Jurkovich GJ, Daranciang E, Dunn CW, Villaveces A, Copass M, Ries RR. Alcohol interventions in a trauma center as a means of reducing the risk of injury recurrence. Ann Surg. 1999 Oct;230(4):473-80; discussion 480-3. doi: 10.1097/00000658-199910000-00003. PMID 10522717
- [Background] Anderson JA, Coscia RL, Cryer HG, et al. Injury does not occur by accident. Resources for the optimal care of the injured patient 2006. Chicago, IL: 2006. p. 115-20.
- [Background] McDonald AJ 3rd, Wang N, Camargo CA Jr. US emergency department visits for alcohol-related diseases and injuries between 1992 and 2000. Arch Intern Med. 2004 Mar 8;164(5):531-7. doi: 10.1001/archinte.164.5.531. PMID 15006830
- [Background] Gentilello LM, Ebel BE, Wickizer TM, Salkever DS, Rivara FP. Alcohol interventions for trauma patients treated in emergency departments and hospitals: a cost benefit analysis. Ann Surg. 2005 Apr;241(4):541-50. doi: 10.1097/01.sla.0000157133.80396.1c. PMID 15798453
- [Background] Wechsler H, Davenport A, Dowdall G, Moeykens B, Castillo S. Health and behavioral consequences of binge drinking in college. A national survey of students at 140 campuses. JAMA. 1994 Dec 7;272(21):1672-7. PMID 7966895
- [Background] Dunn C, Ostafin B. Brief interventions for hospitalized trauma patients. J Trauma. 2005 Sep;59(3 Suppl):S88-93; discussion S94-100. doi: 10.1097/01.ta.0000174682.13138.a3. PMID 16355072
- [Background] Schermer CR. Feasibility of alcohol screening and brief intervention. J Trauma. 2005 Sep;59(3 Suppl):S119-23; discussion S124-33. doi: 10.1097/01.ta.0000174679.12567.7c. PMID 16355047
- [Background] Reboussin BA, Song EY, Shrestha A, Lohman KK, Wolfson M. A latent class analysis of underage problem drinking: evidence from a community sample of 16-20 year olds. Drug Alcohol Depend. 2006 Jul 27;83(3):199-209. doi: 10.1016/j.drugalcdep.2005.11.013. Epub 2005 Dec 15. PMID 16359829
- [Background] Rollnick S. Health Behavior Change: A Guide for paracticioners. New York: Churchill Livingstone; 1999.
- [Background] Cox DR, Oakes DO. Analysis of Survival Data. London: Chapman & Hall; 1984.
- [Background] Tanner MA, Wong WH. Data-based nonparametric estimation of the hazard function with applications to model diagnostics and exploratory analysis. J Am Stat Assoc. 1984; 79:174-182.
- [Background] Andersen P, Gill R. Cox regression model for counting processes: a large sample study. Ann Stat. 1982; 10:1100-1120.
- [Background] Sims DW, Bivins BA, Obeid FN, Horst HM, Sorensen VJ, Fath JJ. Urban trauma: a chronic recurrent disease. J Trauma. 1989 Jul;29(7):940-6; discussion 946-7. PMID 2746704
- [Background] Kaufmann CR, Branas CC, Brawley ML. A population-based study of trauma recidivism. J Trauma. 1998 Aug;45(2):325-31; discussion 331-2. doi: 10.1097/00005373-199808000-00019. PMID 9715190
- [Background] Feuer EJ, Kessler LG. Test statistic and sample size for a two-sample McNemar test. Biometrics. 1989 Jun;45(2):629-36. PMID 2765642
- [Background] Freedman LS. Tables of the number of patients required in clinical trials using the logrank test. Stat Med. 1982 Apr-Jun;1(2):121-9. doi: 10.1002/sim.4780010204. PMID 7187087
- [Background] Collett D. Modeling Survival Data in Medical Research 2003.
- [Background] O'Brien MC, McCoy TP, Champion H, Mitra A, Robbins A, Teuschlser H, Wolfson M, DuRant RH. Single question about drunkenness to detect college students at risk for injury. Acad Emerg Med. 2006 Jun;13(6):629-36. doi: 10.1197/j.aem.2005.12.023. Epub 2006 Apr 13. PMID 16614453